CLINICAL TRIAL: NCT07141719
Title: A Digital Protocol for Neurological Examination Using Eye-Tracking
Brief Title: Collection of Digital Parameters From Parts of the Neurological Examination Using an Eye Tracker
Acronym: NEX-Eye
Status: Not yet recruiting | Type: Observational
Sponsor: University of Kiel (Other)
Responsible Party: Principal Investigator, Walter Maetzler, Prof. Dr. med. Walter Maetzler, University of Kiel
Other Study IDs: D 481/25
Record Dates: First submitted 2025-08-06; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Geriatric; Parkinsons Disease (PD); Progressive Supranuclear Palsy(PSP); Neurological Diseases or Conditions
MeSH Terms: conditions — Parkinson Disease; Supranuclear Palsy, Progressive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Persons with neurological conditions: Patients admitted to the wards and the outpatient clinics of the Department of Neurology, Universitätsklinikum Schleswig-Holstein (UKSH), Campus Kiel

SUMMARY:
The neurological examination (NE) is a cornerstone of clinical neurology, with ocular motor assessment being a key component. Technology offers an opportunity to augment and standardize parts of the NE. Eye-tracking systems provide objective quantitative data on eye movements by continuously tracking the eye over time. This data can be used to derive parameters like saccadic latency, gaze velocity, and fixation stability with a precision that is impossible to achieve through human observation by neurologists. The integration of such technology could enhance the traditional NE.

Before such technology can be widely adopted, its feasibility and acceptability in a clinical population must be established. The primary purpose of this study is to assess the usability of a novel eye-tracking system from the patient's perspective when used in a clinical settings. A secondary purpose is to determine if quantitative data from the eye-tracker correlate with the findings of the traditional clinical neurological examination and to explore whether eye-tracking can provide additional, complementary information not typically captured by standard clinical assessment.

To achieve these aims, the study will assess several outcome measures. The primary outcome measure is the Usability of the Eye-Tracking System, which will be measured using the System Usability Scale (SUS).

Beyond the primary objectives, this study will investigate two secondary objectives.

The first involves assessing the relationship between quantitative eye-tracking parameters and clinical ocular motor assessment. Specifically, the investigators will analyze objective, numerical data obtained from eye-tracking systems and the clinician's subjectively graded assessment of ocular movements derived from the standard neurological examination.

The second is the exploratory analysis of novel eye-tracking biomarkers. This involves quantifying and analyzing eye-tracking parameters not typically assessed during a routine NE. For example, the dynamics of the pupillary light reflex or the frequency of microsaccades. The aim is to identify potential digital biomarkers that could provide additional objective insights into ocular motor function and neurological status.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age.
* Diagnosed or treated for a neurological disease.
* Hospitalized or outpatient of the Department of Neurology, UKSH Campus Kiel.
* Ability of the person to understand oral study information and study information sheet, and willingness to provide a signed and dated informed consent form.

Exclusion criteria:

* Being under legal guardianship
* Impaired decision-making capacity, or temporal or spatial disorientation which may be revealed within ordinary conversation or by a confirmed diagnosis of dementia. In case of doubt, the Montreal Cognitive Assessment (MoCA, pass cutoff score > 18 16) will be administered.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult volunteers hospitalized on the wards and outpatient areas of the Department of Neurology
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
System Usability Scale (SUS) | Baseline (single session, approx. 2-3 hour per participant)
  The System Usability Scale (SUS) is a validated and widely used 10-item questionnaire designed to assess the subjective usability of a system-in this case, a wearable eye-tracking device. Each item is rated on a 5-point Likert scale from Strongly Disagree (1) to Strongly Agree (5).
  The SUS yields a single score ranging from 0 to 100, where higher scores indicate greater perceived usability. A score of 68 is generally considered average; scores above 80 indicate high usability, while scores below 50 suggest usability concerns.
  Usability, in this context, includes perceptions of comfort, system complexity, ease of use, learnability, and willingness to use the system regularly or independently. Participants complete the SUS immediately after using the eye-tracker in a controlled session.

SECONDARY OUTCOMES:
Vestibulo-ocular reflex (VOR) | Baseline (single session, approx. 2-3 hour per participant)
  The vestibulo-ocular reflex (VOR) is measured using the eye-tracker during sitting, standing, and walking. Participants' heads are passively rotated at 100-300 °/s, and the ratio of eye velocity to head velocity (velocity gain) is calculated. A gain of 1.0 indicates perfect VOR function; 0 indicates complete absence.
Vestibulo-ocular reflex suppression (VORS) | Baseline (single session, approx. 2-3 hour per participant)
  Vestibulo-ocular reflex suppression (VORS) is assessed using a head-fixed target. Reflexive eye drift opposite to head movement is measured in sitting, standing, and walking. VORS is calculated as the ratio of eye position to head position (position gain). A score of 100% indicates full expression of the vestibuloocular reflex (VOR) (no suppression), while 0% indicates complete suppression.
Saccades velocity | Baseline (single session, approx. 2-3 hour per participant)
  Saccades are rapid eye movements used to fixate on new visual targets. Using the eye-tracker, saccade velocity (°/s) is recorded and analyzed to detect abnormalities such as slowed or dysmetric movements.
Glabella reflex | Baseline (single session, approx. 2-3 hour per participant)
  The glabellar reflex is assessed by repeated tapping of the participant's glabella. Normally, the blink response habituates after 3-5 taps. Persistent blinking beyond this suggests reduced frontal lobe inhibition. The total number of blinks is recorded.
Pupillary reflex | Baseline (single session, approx. 2-3 hour per participant)
  The pupillary light reflex is assessed by alternately illuminating each eye. An eye-tracker records pupil size, shape, latency, and constriction velocity. Asymmetric responses may indicate neurological deficits. Differences between eyes are quantified, with thresholds based on clinical norms.
Pupil size at rest | Baseline (single session, approx. 2-3 hour per participant)
  Resting pupil size is measured and compared to normative thresholds. Values outside defined ranges are classified as mydriasis (dilated), miosis (constricted), or normal.
Nystagmus at rest, slow phase | Baseline (single session, approx. 2-3 hour per participant)
  Nystagmus is characterized by alternating slow and fast eye movements. At rest, the slow phase velocity (°/s) is recorded during gaze to the left and right using the eye-tracker.
Skew deviation | Baseline (single session, approx. 2-3 hour per participant)
  Skew deviation is assessed using alternate eye cover testing while the participant fixates on a target. A positive result is indicated by vertical correction movements (geotropic/apogeotropic). The presence and magnitude of deviation are evaluated based on predefined thresholds.
Smooth pursuit (SP) number of saccades | Baseline (single session, approx. 2-3 hour per participant)
  Smooth pursuit (SP) is an eye movement in which a moving object is tracked by the eyes without moving the head. The tracking can be saccadic, i.e. jerky, or significantly impaired or incomplete in certain directions, such as upwards. Here, too, the investigators digitally record the extent of the eye movement during neurological examination.
  A disturbance of the SP is indicated by the presence of correction Saccades, which are recorded digitally. As the corrective saccade is a physiological process, the saccade is preceded by a slow phase. During this slow phase, the eye The frequency of the saccades in a time unit is indicated and, if possible, the nature and amplitude. Threshold values for this result from a comparison with the clinical examination and the gestural impression.
  The investigators measure the number of correction saccades per second as a measure of ability to maintain smooth pursuit.
Smooth pursuit (SP) saccade amplitude | Baseline (single session, approx. 2-3 hour per participant)
  The amplitude of the correction saccades, for example in °, during smooth pursuit (SP) also provides information about how saccades can be performed. Together with the number of saccades, it can provide information about the role that the ability to initiate and perform saccades plays during SP. Saccades may play a different role during SP than during gaze shifts.
  The mean amplitude of the saccades is determined.
Smooth pursuit (SP) slow phase velocity | Baseline (single session, approx. 2-3 hour per participant)
  The saccades during smooth pursuit (SP) are preceded by a slow phase, the speed of which can be determined. The investigators calculate the mean of all slow phases in °/s.
Nystagmus at rest, quick phase | Baseline (single session, approx. 2-3 hour per participant)
  Nystagmus is characterized by alternating slow and fast eye movements. The fast phase is expressed as a saccade, which is recorded and measured in degree.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No